CLINICAL TRIAL: NCT03828331
Title: Optimizing Prosthetic and Bicycle Fit for Veterans With Transtibial Amputations
Acronym: BestBikeFit
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: A3010-P
Record Dates: First submitted 2019-01-22; First posted 2019-02-04 (Actual); Results first posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Amputation
Keywords: Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with Transtibial Amputation: The investigators will recruit participants with unilateral transtibial amputations who are at or above a K3 Medicare functional classification level (MFCL), and 18-55 years old. A K3 MFCL means that a person has the ability or potential for ambulation with variable cadence. A person at K3 MFCL is a typical community ambulator who has the ability to traverse most environmental barriers and may have vocational, therapeutic or exercise activity that demands prosthetic use beyond simple locomotion.
  Interventions: Other: Prosthetic/Bicycle Configuration

INTERVENTIONS:
Other: Prosthetic/Bicycle Configuration — The investigators will measure the biomechanics (motion, forces, and muscle activity) and metabolic rates while subjects ride using an initial bike fit and three taller pylon lengths (PL) for the affected leg (AL) in increments of 6.8 mm using a pedal attachment position (PAP) beneath the prosthetic forefoot. Then, using the optimal (most efficient) PL, the investigators will measure the biomechanics and metabolic rates while subjects ride using three shorter crank arm lengths (CALs) for the AL in decrements of 6.8 mm using a PAP beneath the prosthetic forefoot. On Day 2, the investigators will repeat the protocol of Day 1, but have riders use a PAP beneath the pylon for their AL.

SUMMARY:
Bicycling is a promising form of low-impact exercise that could prevent/treat Type 2 diabetes. However, Veterans with transtibial amputations (TTAs) may not effectively utilize bicycling for rehabilitation and exercise due to improper bike fit, socket discomfort, and/or the potential for injury. An optimized prosthetic/bicycle fit could improve comfort and reduce injury risk by decreasing asymmetries between legs, lowering metabolic costs, and improving efficiency for Veterans with TTAs during bicycling. Moreover, the use of objective prosthetic/bicycle fit guidelines would allow clinicians to facilitate shorter appointment times and fewer revisits for Veterans with TTAs. The investigators will determine the physiological and biomechanical effects of different prosthetic and bicycle configurations for Veterans with a TTA to develop optimal prosthetic/bicycle fit guidelines. The investigators hypothesize that a longer prosthetic pylon length and shorter bicycle crank arm length for the affected compared to the unaffected leg along with a pedal attachment position beneath the pylon compared to beneath the forefoot will optimize performance for Veterans with TTAs the investigators' research will integrate evidence-based guidelines to advance rehabilitation and enhance the lives of Veterans with an amputation, thus improving and restoring their function.

DETAILED DESCRIPTION:
Over one million people in the United States have a leg amputation and this number continues to grow due to the prevalence of diabetes and recent military conflicts. Because of the functional impairment caused by an amputation, it is extremely important to advance rehabilitation that optimizes the use of prostheses so that Veterans with amputations can regain the greatest possible level of health, function, and physical activity. Low-impact exercise such as bicycling could facilitate return to work/duty after amputation by improving cardiovascular fitness, muscle strength, endurance, and quality of life for Veterans with transtibial amputations (TTAs). Bicycling as exercise could also prevent the deleterious effects of vascular disease and diabetes by improving cardiovascular function, controlling body weight, decreasing the rate of re-amputation, and improving quality of life for Veterans with TTAs. However, it is likely that discomfort and the increased potential for secondary musculoskeletal injury due to the lack of a proper prosthetic/bike fit discourages Veterans with TTAs from using bicycling for rehabilitation and exercise. Moreover, it is unclear how prosthetic and bicycle components, such as pylon length (PL), pedal attachment position (PAP) beneath the prosthetic forefoot versus the pylon, and crank arm length (CAL) affect the biomechanics, metabolic costs, and comfort/ satisfaction of Veterans with TTAs. Thus, the investigators' goal is to challenge the state-of-the-science by developing evidence-based prosthetic and bicycle fit guidelines that optimize the biomechanics, metabolic costs, efficiency (mechanical power/metabolic power) and comfort/satisfaction for Veterans with TTAs. The Department of Veterans Affairs (VA) and Department of Defense (DoD) Rehabilitation Directive has put forth an initiative that aims to dramatically improve and restore function in wounded Veterans and Service members so that they have the choice to return to active duty or productive civilian employment. The proposed research will establish optimal prosthetic/bicycle fit guidelines, which would enhance function by improving cardiovascular health, controlling body weight, decreasing re-amputation rates, and enhancing quality of life of Veterans with TTAs, thus helping to fulfill this initiative and having high potential impact. Specifically, the investigators aim to: 1) Study 15 Veterans with unilateral TTAs to determine the effects of systematically varying PL, PAP beneath the prosthetic forefoot versus the pylon, and CAL for the affected leg on bicycling biomechanics, metabolic costs, and comfort/satisfaction. 2) Synthesize and disseminate the investigators' findings into practical, evidence-based quantitative prosthetic/bicycle fit guidelines for Veterans with TTAs. The investigators hypothesize that a longer PL and shorter CAL for the affected compared to the unaffected leg along with a PAP beneath the pylon compared to beneath the forefoot will maximize mechanical power symmetry and reduce metabolic cost and muscle activity, and thus maximize efficiency and comfort/satisfaction during bicycling in Veterans with unilateral TTAs. The utilization of evidence-based prosthetic/bicycle fit guidelines that increase symmetry, improve comfort, reduce the risk of injury, decrease metabolic costs, and improve efficiency will directly benefit Veterans with TTAs by increasing their physical activity and function. Optimized prosthetic/bicycle fit guidelines will allow Veterans TTAs who were previously unable to comfortably ride a bicycle, as well as those currently riding a bicycle, to ride longer with less effort and discomfort, potentially leading to an improved quality of life. Moreover, the prosthetic/bicycle fit guidelines generated by this research will ensure that clinicians are able to fit Veterans with TTAs to bicycles more effectively, leading to shorter appointment times and fewer revisits due to enhanced function and reduced comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* One amputation below the knee
* At least 1 year of experience using a prosthesis
* No current problems with the prosthesis or residual limb
* At or above a K3 Medicare Functional Classification Level

Exclusion Criteria:

* Poor general health
* Difficulty with mobility
* Problems with balance or dizziness
* Current serious musculoskeletal injury besides that associated with an amputation
* Cardiovascular, pulmonary, or neurological disease or disorder

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The investigators will recruit 15 subjects with unilateral transtibial amputations from the VA Jewell Clinic, locally, and nationally.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alena Grabowski, PhD BA, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Allen SP, Diaz GB, Grabowski AM. The Effect of Unequal Crank Arm Lengths and Cycling-Specific Prostheses for Recreational Riders with a Transtibial Amputation. Med Sci Sports Exerc. 2024 Oct 1;56(10):1976-1987. doi: 10.1249/MSS.0000000000003480. Epub 2024 May 15. PMID 38768009

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants With Transtibial Amputation
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Transtibial Amputation
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.4 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Mechanical Crank Power Output
Description: The investigators calculated crank power output (W/kg) from the product of pedal torque and velocity and normalized this to participant body mass while participants rode at 1.5 W/kg using different prosthetic and bicycle configurations (pylon length, crank arm length, and pedal attachment position).
Time Frame: Data were collected over 2 days per subject
Measure: Mean (Standard Deviation); unit: W/kg
Groups:
- CSP, AL, 160mm CAL, 0 mm PL; CSP, UL, 160mm CAL, 0 mm PL; CSP, AL, 165mm CAL, 0 mm PL; CSP, UL, 165mm CAL, 0 mm PL; CSP, AL, 170mm CAL, 0 mm PL; CSP, UL, 170mm CAL, 0 mm PL; CSP, AL, 175mm CAL, 0 mm PL; CSP, UL, 175mm CAL, 0 mm PL; CSP, AL, 175mm CAL, 5 mm PL; CSP, UL, 175mm CAL, 5 mm PL; CSP, AL, 175mm CAL, 10 mm PL; CSP, UL, 175mm CAL, 10 mm PL; CSP, AL, 175mm CAL, 15 mm PL; CSP, UL, 175mm CAL, 15 mm PL; DU, AL, 160mm CAL, 0 mm PL; DU, UL, 160mm CAL, 0 mm PL; DU, AL, 165mm CAL, 0 mm PL; DU, UL, 165mm CAL, 0 mm PL; DU, AL, 170mm CAL, 0 mm PL; DU, UL, 170mm CAL, 0 mm PL; DU, AL, 175mm CAL, 0 mm PL; DU, UL, 175mm CAL, 0 mm PL; DU, AL, 175mm CAL, 5 mm PL; DU, UL, 175mm CAL, 5 mm PL; DU, AL, 175mm CAL, 10 mm PL; DU, UL, 175mm CAL, 10 mm PL; DU, AL, 175mm CAL, 15 mm PL; DU, UL, 175mm CAL, 15 mm PL: 12 participants with unilateral transtibial amputation rode using 14 different prosthetic or bicycle configurations where we report data for a cycling-specific prosthesis (CSP) or daily-use prosthesis (DU) for the Affected Leg (AL) or Unaffected Leg (AL) with a given AL crank arm length (CAL) and AL pylon length (PL) reported in mm.
Arm/Group | CSP, AL, 160mm CAL, 0 mm PL | CSP, UL, 160mm CAL, 0 mm PL | CSP, AL, 165mm CAL, 0 mm PL | CSP, UL, 165mm CAL, 0 mm PL | CSP, AL, 170mm CAL, 0 mm PL | CSP, UL, 170mm CAL, 0 mm PL | CSP, AL, 175mm CAL, 0 mm PL | CSP, UL, 175mm CAL, 0 mm PL | CSP, AL, 175mm CAL, 5 mm PL | CSP, UL, 175mm CAL, 5 mm PL | CSP, AL, 175mm CAL, 10 mm PL | CSP, UL, 175mm CAL, 10 mm PL | CSP, AL, 175mm CAL, 15 mm PL | CSP, UL, 175mm CAL, 15 mm PL | DU, AL, 160mm CAL, 0 mm PL | DU, UL, 160mm CAL, 0 mm PL | DU, AL, 165mm CAL, 0 mm PL | DU, UL, 165mm CAL, 0 mm PL | DU, AL, 170mm CAL, 0 mm PL | DU, UL, 170mm CAL, 0 mm PL | DU, AL, 175mm CAL, 0 mm PL | DU, UL, 175mm CAL, 0 mm PL | DU, AL, 175mm CAL, 5 mm PL | DU, UL, 175mm CAL, 5 mm PL | DU, AL, 175mm CAL, 10 mm PL | DU, UL, 175mm CAL, 10 mm PL | DU, AL, 175mm CAL, 15 mm PL | DU, UL, 175mm CAL, 15 mm PL
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
W/kg | 0.59 (0.04) | 0.99 (0.03) | 0.60 (0.04) | 0.97 (0.03) | 0.59 (0.04) | 0.95 (0.03) | 0.60 (0.05) | 0.95 (0.03) | 0.58 (0.04) | 0.98 (0.03) | 0.58 (0.04) | 0.98 (0.03) | 0.57 (0.04) | 0.99 (0.04) | 0.56 (0.04) | 0.98 (0.03) | 0.56 (0.04) | 0.99 (0.03) | 0.56 (0.04) | 0.96 (0.03) | 0.57 (0.04) | 0.97 (0.03) | 0.58 (0.04) | 0.94 (0.03) | 0.56 (0.04) | 0.96 (0.03) | 0.55 (0.05) | 0.99 (0.03)

2. Primary Outcome: Net Metabolic Power
Description: The investigators measured net metabolic power (W/kg) using an equation that considers rates of oxygen consumption and carbon dioxide production and normalized this to participant body mass while participants rode at 1.5 W/kg using different prosthetic and bicycle configurations (pylon length, crank arm length, and pedal attachment position).
Time Frame: Data were collected over 2 days per subject
Measure: Mean (Standard Deviation); unit: W/kg
Groups:
- CSP, 160mm CAL, 0 mm PL; CSP, 165mm CAL, 0 mm PL; CSP, 170mm CAL, 0 mm PL; CSP, 175mm CAL, 0 mm PL; CSP, 175mm CAL, 5 mm PL; CSP, 175mm CAL, 10 mm PL; CSP, 175mm CAL, 15 mm PL; DU, 160mm CAL, 0 mm PL; DU, 165mm CAL, 0 mm PL; DU, 170mm CAL, 0 mm PL; DU, 175mm CAL, 0 mm PL; DU, 175mm CAL, 5 mm PL; DU, 175mm CAL, 10 mm PL; DU, 175mm CAL, 15 mm PL: 12 participants with unilateral transtibial amputation rode using 14 different prosthetic or bicycle configurations where we report data for a cycling-specific prosthesis (CSP) or daily-use prosthesis (DU) with a given affected leg (AL) crank arm length (CAL) and AL pylon length (PL) reported in mm.
Arm/Group | CSP, 160mm CAL, 0 mm PL | CSP, 165mm CAL, 0 mm PL | CSP, 170mm CAL, 0 mm PL | CSP, 175mm CAL, 0 mm PL | CSP, 175mm CAL, 5 mm PL | CSP, 175mm CAL, 10 mm PL | CSP, 175mm CAL, 15 mm PL | DU, 160mm CAL, 0 mm PL | DU, 165mm CAL, 0 mm PL | DU, 170mm CAL, 0 mm PL | DU, 175mm CAL, 0 mm PL | DU, 175mm CAL, 5 mm PL | DU, 175mm CAL, 10 mm PL | DU, 175mm CAL, 15 mm PL
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
W/kg | 7.06 (0.29) | 7.18 (0.30) | 7.09 (0.28) | 6.94 (0.28) | 7.13 (0.30) | 7.14 (0.31) | 7.16 (0.27) | 7.18 (0.28) | 7.19 (0.25) | 7.23 (0.29) | 7.20 (0.27) | 6.74 (0.66) | 7.30 (0.26) | 7.37 (0.28)

3. Primary Outcome: Perceived Comfort (Visual Analog Scale (VAS))
Description: The investigators measured comfort with a questionnaire that has a range of 0-10 that indicates terrible to excellent, respectively, after participants rode at 1.5 W/kg using different prosthetic and bicycle configurations (pylon length, crank arm length, and pedal attachment position).
Time Frame: Data were collected over 2 days per subject
Measure: Mean (Standard Deviation); unit: score on a scale of 0-10
Arm/Group | CSP, 160mm CAL, 0 mm PL | CSP, 165mm CAL, 0 mm PL | CSP, 170mm CAL, 0 mm PL | CSP, 175mm CAL, 0 mm PL | CSP, 175mm CAL, 5 mm PL | CSP, 175mm CAL, 10 mm PL | CSP, 175mm CAL, 15 mm PL | DU, 160mm CAL, 0 mm PL | DU, 165mm CAL, 0 mm PL | DU, 170mm CAL, 0 mm PL | DU, 175mm CAL, 0 mm PL | DU, 175mm CAL, 5 mm PL | DU, 175mm CAL, 10 mm PL | DU, 175mm CAL, 15 mm PL
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
score on a scale of 0-10 | 8.25 (1.42) | 8.08 (1.56) | 8.08 (1.62) | 8.17 (1.53) | 8.17 (1.47) | 8.17 (1.47) | 7.64 (1.57) | 8.42 (1.56) | 8.08 (1.78) | 8.08 (2.15) | 7.67 (2.81) | 7.67 (2.67) | 7.50 (1.73) | 7.00 (1.90)

4. Primary Outcome: Perceived Satisfaction (Prosthesis Evaluation Questionnaire (PEQ))
Description: The investigators measured satisfaction with a questionnaire that has a range of 0-10 that indicates extremely dissatisfied to extremely satisfied, respectively, after participants rode at 1.5 W/kg using different prosthetic and bicycle configurations (pylon length, crank arm length, and pedal attachment position).
Time Frame: Data were collected over 2 days per subject
Measure: Mean (Standard Deviation); unit: score on a scale of 0-10
Arm/Group | CSP, 160mm CAL, 0 mm PL | CSP, 165mm CAL, 0 mm PL | CSP, 170mm CAL, 0 mm PL | CSP, 175mm CAL, 0 mm PL | CSP, 175mm CAL, 5 mm PL | CSP, 175mm CAL, 10 mm PL | CSP, 175mm CAL, 15 mm PL | DU, 160mm CAL, 0 mm PL | DU, 165mm CAL, 0 mm PL | DU, 170mm CAL, 0 mm PL | DU, 175mm CAL, 0 mm PL | DU, 175mm CAL, 5 mm PL | DU, 175mm CAL, 10 mm PL | DU, 175mm CAL, 15 mm PL
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
score on a scale of 0-10 | 7.58 (2.53) | 7.33 (2.64) | 7.17 (2.69) | 7.58 (2.84) | 7.50 (2.68) | 7.33 (2.84) | 6.64 (2.84) | 7.83 (1.85) | 7.75 (2.30) | 7.58 (2.57) | 7.25 (2.60) | 7.42 (2.54) | 7.00 (2.45) | 6.00 (2.72)

ADVERSE EVENTS:
Time Frame: Data were collected over 2 days per participant
Groups:
- Participants With Transtibial Amputation: The investigators will recruit participants with unilateral transtibial amputations who are at or above a K3 Medicare functional classification level (MFCL), and 18-55 years old. A K3 MFCL means that a person has the ability or potential for ambulation with variable cadence. A person at K3 MFCL is a typical community ambulator who has the ability to traverse most environmental barriers and may have vocational, therapeutic or exercise activity that demands prosthetic use beyond simple locomotion.
  Prosthetic/Bicycle Configuration: The investigators will measure the biomechanics (motion and forces) and metabolic rates while subjects ride using an initial bike fit and three taller pylon lengths (PL) for the affected leg (AL) in increments of 6.8 mm using a pedal attachment position (PAP) beneath the prosthetic forefoot. Then, using the optimal (most efficient) PL, the investigators will measure the biomechanics and metabolic rates while subjects ride using three shorter crank arm lengths (CALs) for the AL in decrements of 6.8 mm using a PAP beneath the prosthetic forefoot. On Day 2, the investigators will repeat the protocol of Day 1, but have riders use a PAP beneath the pylon for their AL.
Arm/Group | Participants With Transtibial Amputation
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/31/NCT03828331/Prot_SAP_001.pdf
  • Informed Consent Form (2020-04-27): https://cdn.clinicaltrials.gov/large-docs/31/NCT03828331/ICF_000.pdf